CLINICAL TRIAL: NCT05818228
Title: Reducing Self-Stigma Among Individuals with History of Childhood Maltreatment: a Randomized Controlled Trial
Brief Title: Reducing Self-Stigma Among Individuals with History of Childhood Maltreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Yuval Y Neria, Director of PTSD team at Columbia University, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 8453
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Stigma, Social; Child Abuse; Child Neglect; Help-Seeking Behavior
MeSH Terms: conditions — Social Stigma; Help-Seeking Behavior | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video with Childhood Maltreatment-Related Content (Experimental): Participants will view a video of an actor describing the story of an individual who experienced childhood maltreatment and how they overcame its effects on their life.
  Interventions: Behavioral: Video
- Video without Childhood Maltreatment Content (No Intervention): Participants will view a lifestyle video of an actor describing their day-to-day experiences, without any childhood maltreatment-related themes.

INTERVENTIONS:
Behavioral: Video — A short video aimed at reducing self-stigma among individuals with a history of childhood maltreatment and increasing their help seeking intentions (if needed).
  Arms: Video with Childhood Maltreatment-Related Content

SUMMARY:
Individuals who report experiencing any kind of abuse during childhood report shame and self-blame, often leading to self-stigma and a reluctance to reveal their experiences and seek help. Such stigma may aggravate the mental health consequences of child maltreatment (CM).

The aim of the proposed study is twofold: (1) to evaluate the effectiveness of a brief video-based intervention in reducing self-stigma among individuals who experienced childhood abuse and/or maltreatment, and (2) to increase openness to seeking treatment.

DETAILED DESCRIPTION:
Prior research suggests that social contact-based interventions are the most efficient way of reducing stigma. This study aims to address self-stigma and empower individuals who self-reported experiencing any kind of abuse during childhood and increase their openness to seeking help, if needed.

A total of 1000 adults with self-report experience of any kind of childhood abuse will be recruited to participate in a Randomized Controlled Trial (RCT) testing the efficacy of the intervention. Participants will be randomized into one of two arms: 1) A 2-minute video intervention in which a CM survivor (presented by either a female or male actor) shares their personal CM experience and describes how they were able to overcome feelings of shame and self-blame to seek mental health care; or 2) A 2-minute control video using the same actors, but without CM-related content. Both videos will be preceded by and immediately followed by questionnaires assessing self-stigma and openness to seeking treatment. An additional assessment of emotional engagement will be added immediately following intervention delivery. Following the intervention, there will be a 30-day follow-up to examine potential long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* US resident
* Individuals who endorse yes to one of the following items: physical aggression in family or household, emotional or verbal abuse in family or household, sexual abuse or inappropriate sexual experiences, negligence - physical or emotional, mental illness or substance abuse at home, incarceration of family member
* Fluent in English and able to give informed consent

Exclusion Criteria:

* N/A

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 685 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Self-Stigma Questionnaire - Post-Intervention | Immediately post-intervention
  Change in stigma items from baseline - higher score indicates higher stigma (range of 15 to 60)
Self-Stigma Questionnaire - Follow-Up | 30 days post-intervention
  Change in stigma items from baseline - higher score indicates higher stigma (range of 15 to 60)
Help Seeking Intentions (3 items of the ATSPPH) - Post-Intervention | Immediately post-intervention
  Change in treatment-seeking intentions from baseline - higher score indicates higher help-seeking intentions (range of 3 to 12)
Help Seeking Intentions (3 items of the ATSPPH) - Follow-Up | 30 days post-intervention
  Change in treatment-seeking intentions from baseline - higher score indicates higher help-seeking intentions (range of 3 to 12)

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Neria, PhD, Principal Investigator — NYSPI and Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No